CLINICAL TRIAL: NCT02338297
Title: A Randomized Controlled Trial of Ethanol-gelfoam Mixture(EGM) Versus Gelfoam for the Treatment of Arterioportal Shunts (APS) in Patients With Hepatocellular Carcinoma (HCC) Treated With Transarterial Chemoembolization (TACE)
Brief Title: Therapeutic Effect of Ethanol-gelfoam Mixture for the Treatment of Arterioportal Shunts (APS) in Patients With HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hai-Bin Shi, Director of Radiology Department, the First Affiliated Hospital of Nanjing Medical University, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC001
Record Dates: First submitted 2014-12-18; First posted 2015-01-14 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2015-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; Arterioportal shunts; Transarterial Chemoembolization; Ethanol; Gelfoam; Polyvinyl Alcohol Foam Embolization Particles (PVA)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE+EGM (Experimental): Occlude APS with EGM and perform TACE sequentially
  Interventions: Procedure: TACE; Drug: EGM
- TACE+PVA (Active Comparator): Occlude APS with PVA and perform TACE sequentially
  Interventions: Procedure: TACE; Drug: PVA

INTERVENTIONS:
Procedure: TACE — Transarterial chemoembolisation (TACE)
Drug: EGM — Occlude arterioportal shunts(APS) with ethanol/gelfoam mixture(EGM)
  Arms: TACE+EGM
Drug: PVA — Occlude arterioportal shunts(APS) with PVA
  Arms: TACE+PVA

SUMMARY:
Transcatheter arterial chemoembolization (TACE) is a key palliative treatment for patients with inoperable hepatocellular carcinoma (HCC). Arterioportal shunts (APS) can aggravate portal hypertension and the shunts let lipiodol flow to normal liver tissue and result in poor Lipiodol deposition in the tumor, causing liver ischemia.

Occlusion of APS is a vital and initial step for the following embolization of tumor. Ethanol-gelfoam mixture(EGM) and gelfoam only both can occlude APS in patients with hepatocellular carcinoma (HCC).

The aim of this study was to evaluate the efficacy and safety of EGM in treatment of APS in the procedure of TACE, and to analyze the prognostic factors for survival in this kind of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Child-Pugh A or B cirrhosis
* ECOG performance status Grade 2 or below
* No serious concurrent medical illness
* No prior treatment (including surgery) for HCC
* Histologically or cytologically proven HCC (an alphafetoprotein level > 500 ug/ml in the presence of radiological findings suggestive of HCC in a patient with chronic HBV or HCV infection can be considered eligible at investigator's discretion)
* Unresectable and locally advanced disease without extra-hepatic disease
* Massive expansive or nodular tumor morphology with measurable lesion on CT
* Size of largest tumor <= 15cm in largest dimension
* Number of main tumor <= 5, excluding associated small satellite lesions
* Arterioportal shunts (APS) is found in the angiography of HCC blood supply

Exclusion Criteria:

* History of prior malignancy except skin cancer
* History of significant concurrent medical illness such as ischemic heart disease or heart failure
* History of acute tumor rupture
* Serum creatinine level > 180 umol/L
* Presence of biliary obstruction not amenable to percutaneous drainage
* Child-Pugh C cirrhosis
* History of hepatic encephalopathy, or
* Intractable ascites not controllable by medical therapy, or
* History of variceal bleeding within last 3 months, or
* Serum total bilirubin level > 50 umol/L, or
* Serum albumin level < 28g/L, or
* INR > 1.3
* Presence of extrahepatic metastasis
* Predominantly infiltrative lesion
* Diffuse tumor morphology with extensive lesions involving both lobes.
* Hepatic artery thrombosis, or
* Partial or complete thrombosis of the main portal vein, or
* Tumor invasion of portal branch of contralateral lobe, or
* Hepatic vein tumor thrombus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years
  Defined as time (in days) from time of TACE non-eligibility to death due to any cause, and will be evaluated every 8 weeks in the protocol treatment, and every one year in the follow-up period, respectively. Patients lost to follow-up or alive at the end of the study will be censored at the last date known to be alive.
APS improvement | 2 month
  Changes of Arterioportal Shunts Treated with PVA or EGM

SECONDARY OUTCOMES:
Time To Progression | every 8 weeks, upto 3 years from date of randomization
  Time from randomization to radiological progression. Definition of progression is based on the mRECIST criteria. Deaths during follow-up without evidence of radiological progression are censored.
progression free survival | every 8 weeks, upto 3 years from date of randomization
  Time from randomization to either radiological progression or death. Patients alive and free of progression at the end of follow-up are censored.
Response Rate | every 8 weeks, upto 3 years from date of randomization
  Definition of response is based on the mRECIST criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Shi, MD, PhD., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Zhong da hospital, Southeast university, Nanjing, Jiangsu